CLINICAL TRIAL: NCT03831789
Title: The Neurophysiological Effects of Bilateral Cerebellar rTMS on Cortical Activity and Swallowing Function
Brief Title: The Effects of Bilateral Cerebellar rTMS on Cortical Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRAS 256171
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Dysphagia; Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: All participants over the course of three visits will either have: unilateral cerebellar rTMS or bilateral cerebellar rTMS. However, the order in which they will receive these interventions will be randomly allocated.
Who Masked: Participant
Masking Description: All participants will be masked as to which of the three study arms they have been allocated. All participants over the course of three visits will either have: unilateral cerebellar rTMS or bilateral cerebellar rTMS. However, as specified earlier the order in which they will receive these interventions will be randomly allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral cerebellar rTMS (Active Comparator)
  Interventions: Device: Cerebellar targeted rTMS
- Bilateral cerebellar rTMS (Experimental)
  Interventions: Device: Cerebellar targeted rTMS

INTERVENTIONS:
Device: Cerebellar targeted rTMS — 10 Hz cerebellar rTMS (250 pulses)

SUMMARY:
Swallowing function is controlled by two swallowing centres (one on each half of the brain). There is a dominant and non-dominant swallowing centre. Damage to any part of the brain can lead to swallowing problems, for example in strokes. Recovery of the ability to swallow is associated with increased activity (compensation) over the undamaged centre. The cerebellum is an area of the brain involved in the control and modulation of muscle movements. It is found at the back of the skull.

Over the past few years studies have tried to improve swallowing function using techniques to stimulate regions of the brain and encourage compensation. Repetitive transcranial magnetic stimulation (rTMS) is a technique which can temporarily increase or suppress activity over regions of the brain.

This study will use cerebellar rTMS to attempt to increase activity over the cortical swallowing centres. It will also temporarily suppress activity over the dominant swallowing centre (a virtual lesion) before using cerebellar targeted rTMS to attempt to reverse this suppressive electrical and behavioural effect. The investigators aim to compare the effectiveness of rTMS over the two halves of the cerebellum to rTMS over one half of the cerebellum in increasing activity over the swallowing centres and reversing the suppressive effects of low frequency rTMS 'virtual lesion' over the dominant swallowing centre.

DETAILED DESCRIPTION:
Summary

To determine if 10 Hertz bilateral cerebellar rTMS is more effective than 10 Hertz unilateral cerebellar rTMS or sham in:

1. Increasing PMEP amplitude over the pharyngeal cortical area
2. Reversing focal cortical suppression to the pharyngeal motor cortex induced by a 'virtual lesion'.

This experiment will be performed over six visits to the laboratory.

Experiment Previous studies in our laboratory have shown that focal suppression of the strongest pharyngeal motor representation (1 Hz rTMS for 10 minutes at an intensity of 120% of resting motor threshold) transiently suppresses cortical swallowing activity as measured by PMEP amplitude and function as measured by a swallowing reaction time task, for up to an hour after cessation of rTMS (14, 15). This temporary suppressive effect has been called a cortical 'virtual lesion'. This model has been utilised in several studies (2, 14, 15) as a way of trialling the effects of neurostimulatory interventions in a safe, controlled environment in healthy subjects, before proceeding to patient trials. Studies have also shown that interventions which are capable of reversing the effects of focal cortical suppression more quickly than would ordinarily be the case if the suppressive effects were left to dissipate naturally, are effective in improving post stroke dysphagia (16).

The optimal stimulation sites for the pharyngeal cortical areas and cerebellum will have their resting motor thresholds identified and marked using single pulse TMS with a figure of eight coil (wing diameter of 90mm). Anatomical landmarks will be used to help guide neuronavigation. The vertex of the head will be identified with a tape measure as will the inion (the most prominent part at the back of the skull) (1). Studies have demonstrated that the pharyngeal cortical area is found anterior and lateral to the vertex while both halves of the cerebellum lie inferior and lateral to the inion (1, 15).

Visits 1- 2 (Aim 1 Measurement of Pharyngeal Cortical MEP Amplitude) Cortical and cerebellar PMEPs will be measured by administering single pulse TMS at 10% of stimulator output above resting motor threshold. Ten stimuli (trials) will be given over the pharyngeal motor cortex with greater neuronal activity - lower resting membrane threshold. This stimulus intensity has been shown to give the best reproducibility results for viscerosomatic TMS studies (15). Cerebellar MEPs will be measured by administering 5 stimuli (trials) of single pulse TMS over the cerebellum.

Participants will be randomised to receive one of two cerebellar rTMS interventions (on separate visits):

1. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere (unilateral)
2. Real 10 Hz cerebellar rTMS (250 pulses) to the right and left cerebellar hemispheres (bilateral)

   The effects of the interventions on PMEPs over cortical pharyngeal areas bilaterally will be measured immediately and every fifteen minutes for an hour post intervention. All data will be compared to baseline MEP amplitude.

   Visits 3-4 (Aim 2 Measurement of Pharyngeal Cortical MEP Amplitude after Virtual Lesion) A 'virtual lesion' (1 Hz rTMS for 10 minutes at an intensity of 120% of resting motor threshold) will be administered by holding a figure of eight coil flat over the cortical pharyngeal representation with the highest neurological activity - this is the representation with the lowest resting membrane potential (15). After which, over two visits to the laboratory, unilateral and bilateral cerebellar rTMS will administered to the cerebellar sites identified earlier.

   During these two visits participants will have their baseline pharyngeal MEPs measured in a similar manner to visits 1-2. After focal cortical suppression subjects will be randomised to receive one of two cerebellar rTMS interventions (on separate visits):
3. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere (unilateral)
4. Real 10 Hz cerebellar rTMS (250 pulses) to the right and left cerebellar hemispheres (bilateral)

   The effects of the interventions on PMEPs over cortical pharyngeal areas bilaterally will then be measured immediately and every fifteen minutes for an hour post intervention before being compared to baseline.

   Visits 5-6 (Aim 2 Measurement of Swallowing Accuracy Using Reaction Time Task)

   During these two visits, subjects will have baseline measurements of normal, fast and challenge swallows (*see below for measurement procedure). After focal cortical suppression subjects will be randomised to receive one of two cerebellar rTMS interventions (on separate visits):
5. Real 10 Hz cerebellar rTMS (250 pulses) to the right cerebellar hemisphere (unilateral)
6. Real 10 Hz cerebellar rTMS (250 pulses) to the right and left cerebellar hemispheres (bilateral)

The effects of the interventions on swallowing function will then be measured by repeating normal, fast and challenge swallow reaction times, immediately and at regular intervals for an hour post intervention.

ELIGIBILITY:
Inclusion Criteria:

• Adults above 18 years of age

Exclusion Criteria:

* Epilepsy
* Cardiac pacemaker
* Previous brain surgery
* Previous swallowing problems
* The use of medication which acts on the central nervous system
* Any implanted metal in the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
PMEP | Every 15 minutes for an hour after the intervention.
  Pharyngeal motor evoked potential amplitude (PMEP) amplitude
Swallowing behaviour | Every 15 minutes for an hour after the intervention.
  Swallowing accuracy (number of correct swallows on target out of 10 using a swallowing reaction time task)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, Principal Investigator — University of Manchester
Locations (1):
- Upper G.I laboratory, Salford Royal Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD containing personal identifiable information will not be published. However, anonymised PMEP and swallowing timing data will be published.